CLINICAL TRIAL: NCT04977791
Title: Molecular Landscape of Primary and Acquired Resistance to Immune Checkpoint Inhibitors in Patients With Chinese Advanced Non-small Cell Lung Cancer
Brief Title: Analysis of Drug Resistance in Immune Checkpoint Inhibitors of Non-small Cell Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Xiaomin Niu, Principal Investigator, Shanghai Chest Hospital
Other Study IDs: THORACIC001
Record Dates: First submitted 2021-07-09; First posted 2021-07-27 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer; PD-L1; Resistance; Next-Generation Sequencing
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The specimens are stored in the refrigerator at -20°C or -80°C as specified in the clinical trial protocol. Test specimens and backup specimens should be kept in separate refrigerators to prevent malfunction of one of the refrigerators. Centrifugation time, specimen collection and specimen storage time should be carried out in strict accordance with the requirements of the clinical trial protocol.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Anti-PD-1/PD-L1 monoclonal antibody — Observe a situation before and after immunotherapy
  Other Names: Immune checkpoint inhibitor

SUMMARY:
Immunotherapy has improved the prognosis of non-small cell lung cancer (NSCLC) patients, but about 80% of patients do not respond at all, which is called primary resistance. Absence of the PD-L1 expression is regarded as one of primary resistant reasons to immunotherapy, there are some other reasons which have been reported to be related with the primary resistance, including tumor mutation burden (TMB), microsatellite instability (MSI), tumor neoantigen burden (TNB), HLA genotype, loss of heterozygosity (LOH), intra tumoral heterogeneity (ITH), genome wide doubling (WGD), and ploidy. While some patients initially respond to immunotherapy, later relapse and develop disease progression, which is called acquired resistance, like escaping of interferon signaling pathways or mutations in some important genes such as B2M/JAK1/JAK2.

So the objective of this research is to explore the comprehensive immune molecular markers of primary and acquired resistance to immunotherapy in patients with Chinese advanced NSCLC based on the results of whole exome sequencing (WES) and targeted sequencing (TS)

ELIGIBILITY:
Inclusion Criteria:

* Be able to provide informed consent, and understand and agree to follow the research requirements;
* Advanced non-small cell lung cancer;
* Patients receiving immune checkpoint inhibitor treatment represented by anti-PD-1/PD-L1 monoclonal antibody;
* The patient must be able to provide fresh tumor tissue before- and after- ICIs (50mg of tumor tissue sample/ 2 needles of 18G thick needle puncture) or tumor tissue archived within one year (FFPE tissue block or about 15 pieces [10- 15 sheets] Freshly cut, unstained FFPE slides) and pathology reports (except for advanced non-small cell lung cancer other than neuroendocrine cancer); provide matched 10mL peripheral whole blood samples at the same time;
* ECOG physical fitness status ≤1;
* The patient must have at least one measurable lesion (assessed according to RECIST v1.1);
* Life expectancy ≥ 12 weeks;
* The patient must have adequate organ function, and must be reached absolute neutrophil count (ANC) ≥1.5x10^9/L, platelets ≥100x10^9/L, hemoglobin ≥90g/L, international normalized ratio (INR) or prothrombin time ≤ 1.5x ULN , activated partial thromboplastin time (aPTT)≤1.5x ULN, serum total bilirubin≤1.5x ULN (Patients with Gilbert syndrome can be enrolled if total bilirubin<3x ULN), Aspartate aminotransferase (AST) and alanine aminotransferase (ALT)≤2.5x ULN(Patient with liver metastases, this standard is AST and ALT≤5x ULN) within 7 days before treatment;

Exclusion Criteria:

* Patients with other tumors. Except for basal cell carcinoma of the skin, superficial bladder cancer, squamous cell carcinoma of the skin or cervical cancer in situ, subjects who have received potential radical treatment and have not relapsed within 5 years before the start of treatment can be included in the study;
* Have received any approved systemic anti-tumor immunotherapy before starting the research treatment;
* A history of interstitial lung disease, non-infectious pneumonia or uncontrolled systemic diseases, including diabetes, hypertension, pulmonary fibrosis, acute lung disease, etc.;
* Severe chronic or active infections that require systemic antibacterial, antifungal or antiviral therapy, including tuberculosis infection;
* Known human immunodeficiency virus infection; previous allogeneic stem cell transplantation or organ transplantation;
* The investigator judged that the patient's compliance during the study period was insufficient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese advanced NSCLC patients received immunotherapy who underwent WES and TS sequencing. The investigators studied samples from the patients before- and after- ICIs.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2016-07-21 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 5 years
  The investigator (and the chief radiologist) used the RECIST 1.1 evaluation criteria to evaluate the efficacy indicators. CT or MRI imaging data of the chest and abdomen collected regularly during the screening/baseline period and the study period were used for tumor evaluation. Only when there may be primary or metastatic disease in the pelvis, pelvic imaging is recommended. Any other disease-affected areas (for example, the pelvis and brain) should undergo additional imaging studies based on the individual patient's signs and symptoms. If an unplanned evaluation is performed and it is shown that the patient has not progressed, follow-up evaluation should be performed at the next scheduled visit as much as possible. Scanning/tumor evaluation continued throughout the study period until RECIST 1.1 appeared
Progression-free survival (PFS) | Up to 5 years
  Calculate the time from the immunotherapy to the tumor progression/all-cause death/the end of the follow-up period.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 5 years
  Calculate the time from the immunotherapy to the end of the all-cause death/follow-up period.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiaomin Niu, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Samstein RM, Lee CH, Shoushtari AN, Hellmann MD, Shen R, Janjigian YY, Barron DA, Zehir A, Jordan EJ, Omuro A, Kaley TJ, Kendall SM, Motzer RJ, Hakimi AA, Voss MH, Russo P, Rosenberg J, Iyer G, Bochner BH, Bajorin DF, Al-Ahmadie HA, Chaft JE, Rudin CM, Riely GJ, Baxi S, Ho AL, Wong RJ, Pfister DG, Wolchok JD, Barker CA, Gutin PH, Brennan CW, Tabar V, Mellinghoff IK, DeAngelis LM, Ariyan CE, Lee N, Tap WD, Gounder MM, D'Angelo SP, Saltz L, Stadler ZK, Scher HI, Baselga J, Razavi P, Klebanoff CA, Yaeger R, Segal NH, Ku GY, DeMatteo RP, Ladanyi M, Rizvi NA, Berger MF, Riaz N, Solit DB, Chan TA, Morris LGT. Tumor mutational load predicts survival after immunotherapy across multiple cancer types. Nat Genet. 2019 Feb;51(2):202-206. doi: 10.1038/s41588-018-0312-8. Epub 2019 Jan 14. PMID 30643254
- [Result] Chan TA, Yarchoan M, Jaffee E, Swanton C, Quezada SA, Stenzinger A, Peters S. Development of tumor mutation burden as an immunotherapy biomarker: utility for the oncology clinic. Ann Oncol. 2019 Jan 1;30(1):44-56. doi: 10.1093/annonc/mdy495. PMID 30395155
- [Result] McGranahan N, Furness AJ, Rosenthal R, Ramskov S, Lyngaa R, Saini SK, Jamal-Hanjani M, Wilson GA, Birkbak NJ, Hiley CT, Watkins TB, Shafi S, Murugaesu N, Mitter R, Akarca AU, Linares J, Marafioti T, Henry JY, Van Allen EM, Miao D, Schilling B, Schadendorf D, Garraway LA, Makarov V, Rizvi NA, Snyder A, Hellmann MD, Merghoub T, Wolchok JD, Shukla SA, Wu CJ, Peggs KS, Chan TA, Hadrup SR, Quezada SA, Swanton C. Clonal neoantigens elicit T cell immunoreactivity and sensitivity to immune checkpoint blockade. Science. 2016 Mar 25;351(6280):1463-9. doi: 10.1126/science.aaf1490. Epub 2016 Mar 3. PMID 26940869
- [Result] Chowell D, Morris LGT, Grigg CM, Weber JK, Samstein RM, Makarov V, Kuo F, Kendall SM, Requena D, Riaz N, Greenbaum B, Carroll J, Garon E, Hyman DM, Zehir A, Solit D, Berger M, Zhou R, Rizvi NA, Chan TA. Patient HLA class I genotype influences cancer response to checkpoint blockade immunotherapy. Science. 2018 Feb 2;359(6375):582-587. doi: 10.1126/science.aao4572. Epub 2017 Dec 7. PMID 29217585
- [Result] Klapper JA, Downey SG, Smith FO, Yang JC, Hughes MS, Kammula US, Sherry RM, Royal RE, Steinberg SM, Rosenberg S. High-dose interleukin-2 for the treatment of metastatic renal cell carcinoma : a retrospective analysis of response and survival in patients treated in the surgery branch at the National Cancer Institute between 1986 and 2006. Cancer. 2008 Jul 15;113(2):293-301. doi: 10.1002/cncr.23552. PMID 18457330
- [Result] Remon J, Passiglia F, Ahn MJ, Barlesi F, Forde PM, Garon EB, Gettinger S, Goldberg SB, Herbst RS, Horn L, Kubota K, Lu S, Mezquita L, Paz-Ares L, Popat S, Schalper KA, Skoulidis F, Reck M, Adjei AA, Scagliotti GV. Immune Checkpoint Inhibitors in Thoracic Malignancies: Review of the Existing Evidence by an IASLC Expert Panel and Recommendations. J Thorac Oncol. 2020 Jun;15(6):914-947. doi: 10.1016/j.jtho.2020.03.006. Epub 2020 Mar 14. PMID 32179179